CLINICAL TRIAL: NCT02232750
Title: Evaluation of CPD (Cell Population Data) MNV (Mean Neutrophil Volume) as an Aid in the Diagnosis and Risk Assessment of Sepsis (Protocol # Sepsis 1-14)
Brief Title: Evaluation of CPD MNV as an Aid in the Diagnosis and Risk Assessment of Sepsis (Protocol # Sepsis 1-14)
Acronym: Beckman
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Elliott Crouser MD, Medical Director, Intensive Care Unit, Ohio State University
Other Study IDs: 20141524
Record Dates: First submitted 2014-08-26; First posted 2014-09-05 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Sepsis, Severe Sepsis and Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators hypothesize that CPD parameters will provide improved prediction of sepsis compared to currently employed laboratory parameters. These studies hold the potential to shape practitioner guidelines and improve the timeliness and accuracy with which patients with sepsis are treated today.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 to 90 years)
* Patients presenting to the Emergency Department
* CBC (Complete Blood Count) with differential testing performed and CPD data retrieved

Exclusion Criteria:

* Previously enrolled in this study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Emergency Department
Sampling Method: Probability Sample
Enrollment: 1320 (Actual)
Dates: Start 2014-07-14 (Actual); Primary Completion 2015-08-15 (Actual); Study Completion 2015-08-15 (Actual)

PRIMARY OUTCOMES:
We are measuring CBC (complete blood count) and MNV (Mean Neutrophil Volume) | approximately 10 months
  Evaluate the clinical utility of CPD MNV as an aid in the diagnosis and risk assessment of Emergency Department patients for progression to sepsis, severe sepsis and septic shock.

CONTACTS AND LOCATIONS:
Locations (1):
- Wexner Medical Center at The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Derived] Crouser ED, Parrillo JE, Seymour C, Angus DC, Bicking K, Tejidor L, Magari R, Careaga D, Williams J, Closser DR, Samoszuk M, Herren L, Robart E, Chaves F. Improved Early Detection of Sepsis in the ED With a Novel Monocyte Distribution Width Biomarker. Chest. 2017 Sep;152(3):518-526. doi: 10.1016/j.chest.2017.05.039. Epub 2017 Jun 15. PMID 28625579